CLINICAL TRIAL: NCT03563612
Title: Differential Lung Ventilation vs. CPAP During One Lung Ventilation for Video Assisted Lung Surgery
Brief Title: Differential Lung Ventilation vs. CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr Michal Barak, Senior Anesthesiologist, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RMB-0032-16
Record Dates: First submitted 2018-05-26; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: One Lung Ventilation; Continuous Positive Airway Pressure; Differential Lung Ventilation
Keywords: one lung ventilation; continuous positive airway pressure; differential lung ventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled crossover study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cpap first, differential ventilation later (Active Comparator)
  Interventions: Device: cpap
- differential ventilation first, cpap late (Active Comparator)
  Interventions: Device: cpap

INTERVENTIONS:
Device: cpap — application of cpap to the non-dependent lung, during one lung ventilation

SUMMARY:
In this study we compared the efficacy of continuous positive airway pressure (CPAP) to differential lung ventilation, in terms of patient's oxygenation, during video assisted thoracoscopic lung resection.

DETAILED DESCRIPTION:
Background: One Lung Ventilation (OLV) is the technique used during lung resection surgery in order to facilitate optimal surgical conditions. OLV may result in hypoxemia due to the shunt created. Several techniques are used to overcome the hypoxemia, one of which is continuous positive airway pressure (CPAP) to the non-dependent lung. Another technique is ventilating the non-dependent lung with a minimal volume, thus creating differential lung ventilation (DLV). In this study we compared the efficacy of CPAP to DLV during video assisted thoracoscopic lung resection.

Patients and Method: This is a prospective study of 30 adult patients undergoing elective video assisted thoracoscopic lung lobectomy. Each patient was ventilated in four modes: two lung ventilation, OLV, OLV+CPAP and OLV+DLV. Fifteen patients were ventilated with CPAP first and DLV next, and the other 15 were ventilated with DLV first and then CPAP. Five minutes separated each mode, during which the non-dependent lung was open to room air. We measured the patient's arterial blood gas during each mode of ventilation. The surgeons, who were blinded to the ventilation technique, were asked to assess the surgical conditions at each stage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients diagnised with lung cancer
2. Scheduled to have thoracoscopic lung lobectomy -

Exclusion Criteria:

1. Pregnancy
2. ASA>=4
3. Difficult intubation -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
arterial blood oxygenation | intraoperative
  PaO2

SECONDARY OUTCOMES:
interference with surgical field exposure | intraoperative
  interference
airway pressure in the dependent lung during one lung ventilation | intraoperative
  airway pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Derived] Kremer R, Aboud W, Haberfeld O, Armali M, Barak M. Differential lung ventilation for increased oxygenation during one lung ventilation for video assisted lung surgery. J Cardiothorac Surg. 2019 May 6;14(1):89. doi: 10.1186/s13019-019-0910-2. PMID 31060627